CLINICAL TRIAL: NCT05292859
Title: Long-Term Follow-Up Study for Subjects Enrolled in the Phase I/II Study of Autologous T Cells Using the Sleeping Beauty System to Express T Cell Receptors (TCRs) Reactive Against Cancer-specific Mutations in Subjects With Solid Tumors
Brief Title: Long-Term Follow-up Study of Subjects Treated With Autologous T Cells Using the Sleeping Beauty System to Express TCRs
Status: Completed | Type: Observational
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: TCR001-202
Record Dates: First submitted 2022-02-24; First posted 2022-03-23 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Gynecologic Cancer; Colorectal Cancer; Pancreatic Cancer; Non-small Cell Lung Cancer; Cholangiocarcinoma; Ovarian Cancer; Ovary Neoplasm; Squamous Cell Lung Cancer; Adenocarcinoma of Lung; Adenosquamous Cell Lung Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Cholangiocarcinoma; Ovarian Neoplasms; Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples will be collected for the analysis of TCR-T cell drug product persistence by vector copy number (VCN). The collection of tumor tissue samples is to enable the investigation of changes that may occur within the tumor associated with progression. Tissue samples will be analyzed by NGS (e.g., WES, RNA-Seq, etc.) to evaluate T cell infiltration, TCR-T cell drug product infiltration, presence of HLA alleles and presence of tumor-specific neoantigens. Additional confirmatory analyses of these samples (e.g., immunohistochemistry (IHC) or in situ hybridization (ISH)to verify target expression) may be performed based on emergent data and sufficient sample availability.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rollover subjects from Alaunos Therapeutics TCR-T cell drug product interventional studies: This is a rollover protocol designed to provide long-term follow-up to all subjects previously enrolled in any Alaunos Therapeutics autologous, neoantigen specific TCR-T cell drug product interventional studies.
  Patients will be followed for up to 15 years after dosing of Alaunos Therapeutics autologous, neoantigen specific TCR-T cell drug product.
  Interventions: Biological: Neoantigen specific TCR-T cell drug product

INTERVENTIONS:
Biological: Neoantigen specific TCR-T cell drug product — No study drug is administered in this study. Patients who have received Neoantigen specific TCR-T cell drug product will be evaluated in this trial for long-term safety and efficacy

SUMMARY:
Long-Term Follow-Up Study for Subjects Enrolled in the Phase I/II Study of Autologous T Cells Engineered using the Sleeping Beauty System to Express T cell Receptors (TCRs) Reactive Against Cancer-specific Mutations in Subjects with Solid Tumors

DETAILED DESCRIPTION:
This is a prospective observational, non-interventional study for the long-term follow-up of safety and efficacy for subjects who have received autologous T cells engineered using the Sleeping Beauty System to express T cell receptors (TCRs) reactive against cancer-specific mutations (neoantigen specific TCR-T cells). In this study, subjects will be followed for up to 15 years after initial TCR-T cell drug product administration for evaluation of delayed adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects treated with TCR-T cell drug product on study TCR001-201 or any other Alaunos TCR-T cell drug product study and have either completed their original treatment protocol or have discontinued early.
2. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
3. Subject must be capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
4. Subjects agree to allow clinical samples to be collected and stored at study site and/or Alaunos Therapeutics, Inc. (Alaunos) or designee for testing.

Exclusion Criteria:

1. Subjects that were consented to this LTFU study but did not receive TCR-T cell drug product on study TCR001-201 will be excluded. No other exclusions are permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be enrolled following either the completion or early termination/discontinuation from Study NCT05194735 or any protocol in which patients were administered Neoantigen specific TCR-T cell drug product. Patients will begin the long-term follow-up period regardless of whether they responded to treatment or progressed on treatment. Patients will be followed for up to 15 years post TCR-T cell drug product infusion and will continue to be monitored for safety, immunogenicity and efficacy.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
To assess the long-term safety of subjects that have received neoantigen-specific TCR-T cells | Up to 2 years post TCR-T cell drug product infusion
  Incidence and duration of new related adverse events
To assess the long-term safety of subjects that have received neoantigen-specific TCR-T cells | Up to 15 years post TCR-T cell drug product infusion
  * Incidence and duration of events of special interest, new Serious Adverse Events and new malignancies.
  * Incidence and duration of late onset adverse events
  * Proportion of subjects with adverse events leading to death
  * Incidence of subjects with resolution of adverse events/ serious adverse events and duration of events that began in study TCR001-201 or other clinical trial in which TCR-T cell drug product has been administered.

SECONDARY OUTCOMES:
To investigate translational hypotheses related to TCR-T cell persistence. | Up to 15 years post TCR-T cell drug product infusion
  Duration of TCR-T cell drug product persistence by vector copy number (VCN).
To determine overall survival. | Up to 15 years post TCR-T cell drug product infusion
  Date of TCR-T cell drug product administration to death
To continue the clinical efficacy assessment of TCR-T cell product. | Up to 15 years post TCR-T cell drug product infusion
  Overall response by RECIST 1.1 for subjects who did not have progressive disease on TCR001-201, proportion of subjects receiving subsequent curative therapies
To continue the clinical efficacy assessment of TCR-T cell product. | Up to 15 years post TCR-T cell drug product infusion
  Overall response by iRECIST for subjects who did not have progressive disease on TCR001-201, proportion of subjects receiving subsequent curative therapies
To continue the clinical efficacy assessment of TCR-T cell product. | Up to 15 years post TCR-T cell drug product infusion
  Duration of response (DoR) for subjects who did not have progressive disease on TCR001-201, proportion of subjects receiving subsequent curative therapies
To continue the clinical efficacy assessment of TCR-T cell product. | Up to 15 years post TCR-T cell drug product infusion
  Progression-free survival (PFS) for subjects who did not have progressive disease on TCR001-201, proportion of subjects receiving subsequent curative therapies

OTHER OUTCOMES:
To evaluate the long-term profile of persisting TCR-T cells. | Up to 15 years post TCR-T cell drug product infusion
  Primary and secondary malignancy: presence of TCR-T cells in tumor samples biopsy and autopsy.
To evaluate the long-term profile of persisting TCR-T cells. | Up to 15 years post TCR-T cell drug product infusion
  Determine the TCR-T persistence, defined by the duration of TCR-T cell drug product measurable by vector copy number (VCN) in peripheral blood samples
To evaluate the long-term profile of persisting TCR-T cells. | Up to 15 years post TCR-T cell drug product infusion
  Transposon insertion-site clonality in TCR-T cells over time.
To evaluate the long-term profile of persisting TCR-T cells. | Up to 15 years post TCR-T cell drug product infusion
  To evaluate changes in T cell infiltration that may occur within the tumor associated with disease progression following TCR-T cell infusion
To evaluate the long-term profile of persisting TCR-T cells. | Up to 15 years post TCR-T cell drug product infusion
  To evaluate infiltration of TCR-T cells within tumor tissue following disease progression
To evaluate the long-term profile of persisting TCR-T cells. | Up to 15 years post TCR-T cell drug product infusion
  To evaluate the presence of HLA alleles within the tumor associated with disease progression following TCR-T cell infusion
To evaluate the long-term profile of persisting TCR-T cells. | Up to 15 years post TCR-T cell drug product infusion
  To evaluate changes in the presence of tumor-specific neoantigens within the tumor associated with disease progression following TCR-T cell infusion

CONTACTS AND LOCATIONS:
Overall Officials: Scott Kopetz, MD, PhD, Principal Investigator — MD Anderson
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States